CLINICAL TRIAL: NCT01234831
Title: A Novel Approach to MRSA Screening of Colonized Patients and Impact on Hospital Resource Allocation and Patient Care
Brief Title: A Novel Approach to Methicillin-resistant Staphylococcus Aureus (MRSA) Screening of Colonized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Erica S. Shenoy, Assistant Chief, Infection Control Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010P001336
Record Dates: First submitted 2010-10-28; First posted 2010-11-04 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-09

CONDITIONS: MRSA Colonization
Keywords: MRSA; colonization; nucleic acid amplification; chromogenic agar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Screening (Other): Patients randomized to active screening will have two nasal swabs collected daily for 3 days, for both nucleic acid amplification and culture (CHROMagar)assays.
  Interventions: Device: nucleic acid amplification of nasal swab; nasal swab culture
- Passive Screening (Other): Patients randomized to passive screening will not actively be identified for testing but may be tested using culture-based algorithm by care team.
  Interventions: Other: Nasal swab culture

INTERVENTIONS:
Device: nucleic acid amplification of nasal swab; nasal swab culture — Nasal swab is performed and analyzed using nucleic acid amplification to determine the presence or absence of MRSA DNA. One nasal swab is performed each day for three consecutive days during hospitalization.
  Other Names: Cepheid Xpert MRSA; BD CHROMagar
  Arms: Active Screening
Other: Nasal swab culture — Nasal swabs are obtained if the clinician caring for the patient identifies the patient as eligible to be screened for colonization. An algorithm for screening eligible patients is available electronically as part of the patient's standard medical record to the clinicians providing care.
  Other Names: BD CHROMagar
  Arms: Passive Screening

SUMMARY:
Methicillin-resistant Staphylococcus aureus (MRSA) is endemic in hospital settings. Colonization with MRSA puts patients at increased risk for invasive infections, and MRSA infections have been associated with high costs and adverse clinic outcomes. Patients can clear MRSA spontaneously. Improved approaches for identifying patients who are no longer colonized are needed; we hypothesize that more sensitive nucleic acid amplification can be used to improve identification of patients who are no longer colonized.

DETAILED DESCRIPTION:
Compared with patients with methicillin-susceptible Staphylococcus aureus (MSSA) bacteremia, patients with MRSA bacteremia remained in the hospital for two more days on average and had a median attributable increment in hospital charges of approximately $7000.

MRSA status is a determinant of bed allocation, especially in shared-room settings, which represent the most common organization in the US and globally. Based on guidelines from the Centers for Disease Control and Prevention, once patients are designated as having had a positive MRSA culture (either colonized or from a clinical isolate), they require Contact Precautions. This requirement translates into either cohorting with other patients with similar precautions status (i.e., two patients with MRSA share a room) or placement in a private room in the hospital. Cohorting is not the preferred infection control method, but in shared-room settings, it is the most common scenario, particularly in hospitals with high occupancy.

Individuals can clear MRSA colonization spontaneously. In fact, up to 38% of patients with MRSA-positive cultures taken greater than 3 months prior were found to be MRSA-negative during a re-screening program conducted by the Massachusetts General Hospital Infection Control Unit from 2004-2006. Other studies have demonstrated that a majority of patients are likely to clear colonization at various time points from original documentation of MRSA infection or colonization. There is currently no standardized approach or accepted guidelines for addressing screening for clearance of colonization in the growing pool of patients who have previous MRSA colonization/infection. Many organizations do provide guidelines for screening, but these guidelines are not based on rigorous study, have a variety of permutations, and have neither consensus acceptance nor adequate implementation among the medical community.

The status quo limits bed availability and delays patient discharge to rehabilitation facilities, adversely affecting quality and efficiency, and resulting in use of additional hospital resources. In addition to problems associated with patient flow for admissions and discharges, precaution status results in additional disruptions of patient care through "bed moves" to accommodate the use of shared rooms by like patients needing Contact Precautions.

A patient's precaution status affects his/her care from admission through discharge. During pre-admission, patients identified as previously having MRSA are affected by bed shortages and delays to admission while in emergency departments. While admitted, under current practices, patients who have in fact cleared MRSA may be cohorted with those who have active infection or persistent colonization, putting them at risk of recolonization and hospital acquired infection (HAI). Finally, patients who are on precautions for MRSA often have delayed discharge to rehabilitation or nursing facilities because of bed constraints similar to those experienced by acute care facilities.

We hypothesize that the use of more sensitive Polymerase Chain Reaction (PCR) methods detecting MRSA in nasal swabs can facilitate identification of true negative patients and can reliably do so with a single negative test in a shorter period of time, thereby greatly facilitating the ability to complete testing on a larger proportion of patients.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* last positive MRSA culture greater than 3 months old
* admitted to hospital

Exclusion Criteria:

* age < 18
* last positive MRSA culture less than or equal to 3 months old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Hooper, MD, Principal Investigator — Massachusetts General Hospital; Erica S Shenoy, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Shenoy ES, Noubary F, Kim J, Rosenberg ES, Cotter JA, Lee H, Walensky RP, Hooper DC. Concordance of PCR and culture from nasal swabs for detection of methicillin-resistant Staphylococcus aureus in a setting of concurrent antistaphylococcal antibiotics. J Clin Microbiol. 2014 Apr;52(4):1235-7. doi: 10.1128/JCM.02972-13. Epub 2014 Jan 22. PMID 24452168
- [Derived] Shenoy ES, Kim J, Rosenberg ES, Cotter JA, Lee H, Walensky RP, Hooper DC. Discontinuation of contact precautions for methicillin-resistant staphylococcus aureus: a randomized controlled trial comparing passive and active screening with culture and polymerase chain reaction. Clin Infect Dis. 2013 Jul;57(2):176-84. doi: 10.1093/cid/cit206. Epub 2013 Apr 9. PMID 23572482
- See also: Clin Infect Dis 2013 May 10. [Epub ahead of print] — http://www.ncbi.nlm.nih.gov/pubmed/23572482
- See also: J Clin Microbiol. 2014 Apr;52(4):1235-7. doi: 10.1128/JCM.02972-13. Epub 2014 Jan 22. — http://www.ncbi.nlm.nih.gov/pubmed/24452168

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Screening | Passive Screening
Started | 261 | 202
Completed | 259 | 198
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Screening | Passive Screening | Total
Number analyzed (Participants) | 261 | 202 | 463
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 96 | 222
  >=65 years | 135 | 106 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (16.77) | 62.9 (18.45) | 63.47 (17.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 86 | 177
  Male | 170 | 116 | 286
Region of Enrollment [Number; unit: participants]
  United States | 261 | 202 | 463

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Single Negative Polymerase Chain Reaction (PCR) Result and 3 Negative Culture Assays
Description: This outcome is the negative predictive value of a single PCR assay for subjects with a history of prior MRSA infection or colonization.
Time Frame: 1 year
Population: Only patients randomized to the Active Screening arm who had 3 pairs of completed nasal swabs could be analyzed for this outcome measure which is the negative predictive value of the first PCR sample compared to three culture samples for subjects with a history of prior MRSA infection or colonization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Active Screening: Patients randomized to the Active Screening arm will have paired nasal swabs collected daily for 3 days; one processed using nucleic acid amplification and the other using culture (CHROMagar) assays.
Arm/Group | Active Screening
Number analyzed (Participants) | 191
percentage of participants | 96.6 [91.6 to 99.1]

2. Primary Outcome: Completion of Screening Protocol in Both Trial Arms
Description: Rate at which subjects in both trial arms complete the 3-swab protocol.
Time Frame: 1 year
Population: Participants in both the Active Screening arm and Passive Screening arm who completed the 3-swab protocol.
Measure: Number; unit: percentage of subjects completed 3 swabs
Groups:
- Passive Screening: Patients randomized to the Passive Screening arm will not actively be identified for testing but may be tested using institutional culture-based protocol available to all primary care teams.
Arm/Group | Active Screening | Passive Screening
Number analyzed (Participants) | 259 | 198
percentage of subjects completed 3 swabs | 73.7 | 9.6

3. Primary Outcome: Discontinuation of Contact Precautions in Both Trial Arms
Description: Patients known to have MRSA require Contact Precautions based on current recommendations from the Center for Disease Control and Prevention (CDC). Contact Precautions mean that hospitalized patients with a history of MRSA infection or colonization are isolated in a private room or together with patients who have the same Contact Precautions status (i.e. both with MRSA). Healthcare workers caring for such patients must wear protective gowns and gloves during interactions and use of equipment dedicated to that patient is recommended. For this study, "Contact Precautions are discontinued" refers to the practice of discontinuation of Contact Precautions once subjects meet criteria based on institutional infection control policy: history of MRSA but no positive culture in preceding 90 days and three negative nasal surveillance cultures obtained at least 24 hours apart in the absence of concurrent antibiotic use.
Time Frame: 1 year
Population: Analysis was performed on patients in both the Active Screening arm and Passive Screening arm who had completed the 3-swab protocol and all 3 swabs were negative.
Measure: Number; unit: percentage of MRSA CP discontinued
Arm/Group | Active Screening | Passive Screening
Number analyzed (Participants) | 125 | 15
percentage of MRSA CP discontinued | 55.2 | 86.7

4. Secondary Outcome: Number of Subjects With a Single Positive PCR Result and at Least 1 Positive Culture Assay
Description: This outcome is the positive predictive value of a single PCR assay for subjects with a history of prior MRSA infection or colonization who completed the 3 swab protocol.
Time Frame: 1 year
Population: Number of participants in the Active Screening arm who had completed the 3-swab protocol.
Measure: Number; unit: participants
Arm/Group | Active Screening
Number analyzed (Participants) | 191
participants | 62

5. Secondary Outcome: Sensitivity of First PCR Assay
Description: Sensitivity of the first PCR assay for subjects enrolled in active arm of trial.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Arm/Group | Active Screening
Number analyzed (Participants) | 191
percentage of true positives | 93.9 [85.4 to 97.6]

6. Secondary Outcome: Specificity of First PCR Assay.
Description: Specificity of the first PCR assay for subjects enrolled in active arm of trial.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of true negatives
Arm/Group | Active Screening
Number analyzed (Participants) | 191
percentage of true negatives | 92.0 [85.9 to 95.6]

7. Secondary Outcome: Rate of Recolonization or Documented Infection With MRSA
Description: Prospective review of microbiological data for patients enrolled in the trial to determine rate of recolonization or documented infection. Subjects in the Intervention Arm of the study who had documented clearance of colonization and met criteria for discontinuation of contract precautions, and had CP discontinued by staff (N=69) were included. Subjects who had a visit at MGH through 12/31/2012 during which a microbiology sample was obtained and MRSA was recovered (clinical or surveillance) were included.
Time Frame: 2 years
Population: We reviewed the data on the 69 subjects who were enrolled in the intervention arm of the trial who were cleared of colonization based on the study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Active Screening With Contact Precautions Removed: Patients randomized to active screening will have two nasal swabs collected daily for 3 days, for both nucleic acid amplification and culture (CHROMagar)assays. Contact Precautions will be removed for subjects who are cleared of colonization based on the study intervention.
Arm/Group | Active Screening With Contact Precautions Removed
Number analyzed (Participants) | 69
Participants | 8

ADVERSE EVENTS:
Arm/Group | Active Screening
Serious Adverse Events (participants affected / at risk) | 0/463
Other Adverse Events (participants affected / at risk) | 0/463

LIMITATIONS AND CAVEATS:
This study was conducted at a single tertiary academic center and in the absence of any national guidelines, we implemented the local standard of care for discontinuation of CP, the components of which are found in variable combinations nationally.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No